CLINICAL TRIAL: NCT05937789
Title: Effects of Early Vitamin D3 Supplementation on Clinical Outcomes for Critically Ill Patients
Brief Title: Early Vitamin D3 Supplementation for Critically Ill Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 202305074RIPC
Record Dates: First submitted 2023-06-30; First posted 2023-07-10 (Actual); Last update posted 2024-08-16 (Actual); Status verified 2024-07

CONDITIONS: Vitamin D Deficiency; Critical Illness
Keywords: vitamin D; calcidiol levels; critically ill
MeSH Terms: conditions — Vitamin D Deficiency; Critical Illness | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Control1 (Placebo Comparator): Participants with serum 25(OH)D levels of 15-19.9 ng/mL, receiving 40 cc. medium-chain triglyceride (MCT) supplement.
  Interventions: Dietary Supplement: Medium Chain Triglycerides (MCT)
- Control2 (Placebo Comparator): Participants with serum 25(OH)D levels of 12-14.9 ng/mL, receiving 50 cc. MCT supplement.
  Interventions: Dietary Supplement: Medium Chain Triglycerides (MCT)
- Control3 (Placebo Comparator): Participants with serum 25(OH)D levels below 12 ng/mL, receiving 60 cc. MCT supplement.
  Interventions: Dietary Supplement: Medium Chain Triglycerides (MCT)
- Vitamin D1 (Experimental): Participants with serum 25(OH)D levels of 15-19.9 ng/mL, receiving vitamin D3 of 576,000 IU supplement
  Interventions: Dietary Supplement: Vitamin D3
- Vitamin D2 (Experimental): Participants with serum 25(OH)D levels of 12-14.9 ng/mL, receiving vitamin D3 of 720,000 IU supplement
  Interventions: Dietary Supplement: Vitamin D3
- Vitamin D3 (Experimental): Participants with serum 25(OH)D levels below 12 ng/mL, receiving vitamin D3 of 864,000 IU supplement
  Interventions: Dietary Supplement: Vitamin D3

INTERVENTIONS:
Dietary Supplement: Vitamin D3 — Dose of vitamin D3 depends on participant's serum 25(OH)D levels, with one sample bottle contains 72,000 IU of vitamin D3; Intervention starts on ICU day 3 with a frequency of 1 ampule every 3 hours and is completed within the following 48 hours
  Arms: Vitamin D1; Vitamin D2; Vitamin D3
Dietary Supplement: Medium Chain Triglycerides (MCT) — Dose of MCT depends on participant's serum 25(OH)D levels, with one sample bottle contains 5 cc. of MCT; Intervention starts on ICU day 3 with a frequency of 1 ampule every 3 hours and is completed within the following 48 hours
  Arms: Control1; Control2; Control3

SUMMARY:
There are no clear international guidelines for dosing vitamin D based on deficiency severity. Therefore, a new clinical trial is needed to evaluate the benefits of early vitamin D supplementation in maintaining sufficient levels for critically ill patients. The investigators conducted a multicenter clinical trial in Taiwan focusing on vitamin D and critically ill patients. 240 patients with low calcidiol levels will be enrolled and be provided varying supplementation doses to maintain their serum calcidiol levels ≥ 30 ng/mL within 30 days of ICU admission. The serum levels of calcidiol and PTH will be measured on Day 0, Day 7, Day 14 and Day 30 before and after vitamin D supplementation. The results will serve as a valuable reference for intensivists when formulating appropriate vitamin D treatment strategy to maximize clinical benefits for critically ill patients.

DETAILED DESCRIPTION:
Recent studies have highlighted a prevalent vitamin D deficiency in critically ill patients, ranging from 26% to 82%. These patients experience longer ICU stays, higher medical expenses, and increased sepsis-related mortality. The investigators conducted a multicenter clinical trial in Taiwan focusing on vitamin D and critically ill patients. In the first phase, the epidemiological investigation found significantly lower serum calcidiol levels of approximately 20.9 ng/mL compared to the normal range of 30-60 ng/mL in ICU patients. The second phase, a randomized control study, preliminarily demonstrated that supplementing 576,000 IU of vitamin D3 in critically ill patients with serum calcidiol levels below 20 ng/mL significantly reduced the risk of multidrug resistant bacterial infections within 30 days. An Austrian trial also showed that adequate vitamin D supplementation lowered in-hospital mortality in severely deficient patients. The importance of vitamin D supplementation for critically ill patients with vitamin D deficiency is evident, as their clinical prognosis is closely related to achieving adequate serum calcidiol levels. However, there are no clear international guidelines for dosing vitamin D based on deficiency severity. Therefore, a new clinical trial is needed to evaluate the benefits of early vitamin D supplementation in maintaining sufficient levels for critically ill patients. The investigators will enroll 240 patients with low calcidiol levels and provide varying supplementation doses to maintain their serum calcidiol levels ≥ 30 ng/mL within 30 days of ICU admission. The serum levels of calcidiol and PTH will be measured on Day 0, Day 7, Day 14 and Day 30 before and after vitamin D supplementation. The results will serve as a valuable reference for intensivists when formulating appropriate vitamin D treatment strategy to maximize clinical benefits for critically ill patients.

ELIGIBILITY:
Inclusion Criteria:

* ≥18-year-old critically ill patient.
* ICU admission < 24 hours.
* Baseline 25(OH)D levels within 24 hours of ICU admission < 20 ng/mL.
* Expected ICU length of stay ≥ 72 hours.

Exclusion Criteria:

* Hypercalcemia (ie. total serum calcium levels > 2.6 mmol/L).
* Disorders affecting serum 25(OH)D levels, calcium metabolism, or bone metabolism (eg, parathyroid disease, rickets, or severe cirrhosis [Child C]).
* Having received high-dose vitamin D3 therapy (ie. > 2,000 IU daily or a single dose of ≥ 10,000 IU) within the past four weeks.
* Active COVID-19 at ICU admission.
* Organ transplant.
* Having had tuberculosis, sarcoidosis or kidney stones within the past year.
* Having renal dialysis, continuous kidney replacement therapy (CKRT), acute kidney injury (AKI).
* Having ICU admission within the past three months.
* Non-native-speaking patients and their families
* Pregnant women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2024-01-22 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
30-day mortality rate | 30 days
  30-day mortality rate after intervention with the study samples.

SECONDARY OUTCOMES:
30-day mortality rate of patients who survives >7 days | 30 days
  30-day mortality rate of patients who survives >7 days after intervention with the study. samples
Length of ICU stay for surviving patients | 30 days
  Length of ICU stay for surviving patients.
Length of hospital stay for surviving patients | 30 days
  Length of hospital stay for surviving patients.
30-day mortality based on serum 25(OH)D levels on day 7 | 30 days
  Comparison of 30-day mortality between the two treatment groups based on serum 25(OH)D levels on day 7: ≥ 30 ng/mL vs. < 30 ng/mL.
30-day mortality based on serum 25(OH)D levels on day 30 | 30 days
  Comparison of 30-day mortality between the two treatment groups based on serum 25(OH)D levels on day 30: ≥ 30 ng/mL vs. < 30 ng/mL.
30-day mortality based on APACHE II scores at ICU 24 hours | 30 days
  Comparison of 30-day mortality between the three groups based on 24-hour APACHE II scores: <20, 20-39, and ≥39.
Correlation of 25(OH)D increment after vitamin D supplement and body weight | 7 days
  Correlation between 25(OH)D levels and body weight on day 7 after supplementation in the treatment group.

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No